CLINICAL TRIAL: NCT06417866
Title: Enhancing Informed Consent Utilizing a Spinal Model for Lumbar Epidural Steroid Injection: A Prospective Randomized Controlled Study.
Brief Title: Informed Consent Using a Spinal Model
Status: Completed | Type: Observational
Sponsor: Ankara University (Other)
Responsible Party: Principal Investigator, Hanzade Aybuke Unal, Medical Doctor, Ankara University
Other Study IDs: 2023/719
Record Dates: First submitted 2024-05-10; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Anxiety; Depression; Pain
Keywords: pain; anxiety
MeSH Terms: conditions — Anxiety Disorders; Depression; Pain | interventions — Informed Consent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- standard informed consent: standard verbal and written informed consent form
  Interventions: Other: informed consent
- visual spinal model: standard verbal and written informed consent form + visual spinal model
  Interventions: Other: spine model

INTERVENTIONS:
Other: informed consent — standard verbal and written informed consent
  Groups: standard informed consent
Other: spine model — standard verbal and written informed consent + visual spine model
  Groups: visual spinal model

SUMMARY:
Informed consent is the first step in every medical procedure. It is important for the patient to clearly understand how the procedure will be performed, what to expect from the process, and the possible complications. Any of the specified processes disruption may alter procedure satisfaction and treatment outcomes. Studies have reported that providing insufficient information before interventional procedures increases anxiety and the severity of pain during the procedure. In this study, alongside the standard procedures for obtaining oral and written consent, it is envisaged to augment patient comprehension and engagement by visually demonstrating the treatment areas and needle insertion points using a spinal model. Within the study framework, patients will be presented with both verbal and written informed consent, supplemented by visual aids utilizing a spinal model. The study aims to assess and compare the efficacy of this enhanced consent process in terms of patient understanding, procedural acceptance, and subsequent satisfaction levels.

DETAILED DESCRIPTION:
The informed consent process includes the processes of explanation, understanding, selection and approval of the volunteer. For informed consent to be valid, the patient must obtain sufficient information about the procedure, be in communication with the physician, be voluntary, and have the capacity to give consent. In our country, informed consent forms usually include a physician-patient interview, reading and signing of the written text. Although informed consent forms are written in a language that patients can understand, they can be complicated for patients. Studies have shown that video and other audio-visual materials significantly improve patients' understanding of the subject. It has been proven to facilitate follow-up and increase compliance with the treatment plan. Informed consent using multimedia tools is reported to be effective.

Lumbar radiculopathy is a condition characterized by pain that can affect daily life and is one of the most common causes of low back pain. Epidural steroid injections can be applied to patients that do not benefit from conservative treatment. Lumbar epidural steroid injections are a minimally invasive procedure and their method of application in society is not clearly known. This procedure is performed with a needle and accompanied by imaging techniques, without any incision. There are a limited number of studies on informed consent forms before lumbar epidural applications. In a study, it was found that patients who did not understand the consent form or received insufficient information had lower post-procedure satisfaction. In another study it stated that in patients who were given a brochure explaining the procedure in addition to verbal and written consent, giving the brochure had no effect on pre-procedure anxiety and post-procedure pain severity.

Verbal and written consent is routinely obtained from patients who are planned to receive lumbar epidural steroid injection in our clinic. In this study, in addition to the routine oral and written consent, it is planned to show the patients the areas to be treated and where the needle will be placed via a spinal model. Within the scope of the study, patients were provided with verbal and written informed consent and visual illustrations through a spine model in addition to verbal and written informed consent. The aim of the study is to compare the level of understanding of consent, acceptance of the procedure and its effect on patient satisfaction after the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for lumbar epidural steroid injection due to radicular pain
* Patients who gave consent to participate in the study

Exclusion Criteria:

* Presence of psychiatric illness that is unstable/not controlled by medical treatment
* Pregnant patients
* Patients who have previously received epidural steroid injections
* Patients who did not give consent to participate in the study
* Patients with cognitive impairment
* Patients with major coagulopathy
* Patients with mental disabilities
* Illiterate patients

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients between the ages of 18 and 65 who are scheduled to receive lumbar epidural steroid injection due to radicular pain will be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 168 (Actual)
Dates: Start 2024-01-02 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Informed consent form comprehension assessment | 1 day
  The degree of understanding of the informed consent form evaluation with a 3-point Likert scale.
Patient satisfaction after the procedure | 1st hour
  The degree of patient satisfaction evaluation after the lumbar epidural steroid injection with a 5-point Likert scale.
anxiety and depression | 1 day
  anxiety and depression evaluation before the procedure with Hospital Anxiety and Depression Scale (HADS). A score of 0-7 in the survey indicates normal, 8-10 points indicates borderline, and 11 and above indicates anxiety/depression.The maximum score that can be obtained from the survey is 42, and higher scores are associated with worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Hanzade A Unal, MD, Study Director — Ankara University
Locations (1):
- Ankara University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ketelaars PJW, Buskes MHM, Bosgraaf RP, van Hamont D, Prins JB, Massuger LFAG, Melchers WJG, Bekkers RLM. The effect of video information on anxiety levels in women attending colposcopy: a randomized controlled trial. Acta Oncol. 2017 Dec;56(12):1728-1733. doi: 10.1080/0284186X.2017.1355108. Epub 2017 Aug 1. PMID 28760058
- [Background] Bahar Ozdemir Y, Sencan S, Ercalik T, Kokar S, Gunduz OH. Do informative leaflets affect pre-procedural anxiety and immediate pain after transforaminal epidural steroid injections? A prospective randomized controlled study. Agri. 2021 Jan;33(1):1-6. doi: 10.14744/agri.2020.27048. PMID 34254651